CLINICAL TRIAL: NCT01289223
Title: A Randomised, Open Label, Multi-centre, Phase III Study to Investigate the Efficacy of Bendamustine Compared to Treatment of Physician's Choice in the Treatment of Subjects With Indolent Non-Hodgkin's Lymphoma (NHL) Refractory to Rituximab
Brief Title: A Trial to Investigate the Efficacy of Bendamustine in Patients With Indolent Non-Hodgkin's Lymphoma (NHL) Refractory to Rituximab.
Acronym: ROBIN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Ongoing challenges to successfully recruit the required number of subjects
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BDM3502; 2010-022102-41 (EudraCT Number)
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Indolent B-cell NHL
Keywords: Indolent B-cell NHL, bendamustine, rituximab, progression-free survival

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment of Physicians Choice (Active Comparator): Defined as any cancer specific therapy or best supportive care. Treatment should be given according to the label and based upon local institutional medical practice and clinical judgement.
  Interventions: Other: Treatment of Physicians Choice
- Bendamustine IV (Experimental): Up to 8 cycles of Bendamustine (120mg/m2 Days 1 and 2, every 21 days (+ 3 days).
  Interventions: Drug: Bendamustine IV

INTERVENTIONS:
Drug: Bendamustine IV
  Arms: Bendamustine IV
Other: Treatment of Physicians Choice — Defined as any cancer specific therapy or best supportive care. Treatment should be given according to the label and based upon local institutional medical practice and clinical judgement.
  Other Names: Defined as any cancer specific therapy or best supportive care.
  Arms: Treatment of Physicians Choice

SUMMARY:
To compare the efficacy of bendamustine against treatment of physician's choice on progression-free survival in subjects with indolent B-cell NHL.

DETAILED DESCRIPTION:
To test whether bendamustine will improve progression-free survival in subjects with indolent B-cell NHL that did not respond (stable disease or progressive disease) to rituximab or a rituximab-containing regimen during or within 6 months of the last rituximab treatment compared to treatment of physican's choice.

ELIGIBILITY:
Inclusion Criteria:

1. Indolent B-cell lymphoma: grades 1-3a follicular, small lymphocytic, lymphoplasmacytic, and marginal zone lymphoma; stages III-IV, or bulky disease stage II (i.e. as any single mass > 5 cm in any direction) defined according to WHO Classification, 2008
2. CT imaging in screening phase (based on local evaluation) showing 2 or more clearly demarcated lesions with a largest diameter ≥ 1.5 cm, or 1 clearly demarcated lesion with a largest diameter ≥ 2.0 cm. CT imaging performed at screening will be considered the baseline image
3. Indolent B-cell NHL that remains stable or unresponsive during or within 6 months of treatment with rituximab or a rituximab-containing regimen:

   * Maintaining stable disease or failure to achieve PR to rituximab-based therapy. (CT imaging will support this finding, and will be performed at least 30 days after the last dose of rituximab-based therapy) or,
   * Disease progression while on rituximab-based therapy (e.g., includes 4 weekly courses of rituximab given at 6 week intervals) or,
   * Disease progression in subjects with stable disease or better response to rituximab-based therapy < 6 months of the last dose of rituximab Note: Subjects must have received at least 4 infusions of rituximab (either as monotherapy or in combination with any chemotherapy).
4. Screening laboratory values:

   * Platelets ≥ 75,000/µL (7 x 109 cells/L)
   * Absolute neutrophil count (ANC) ≥ 1,000/µL (1.0 x 109 cells/L)
   * ALT, AST and alkaline phosphatase ≤ 2.5 ULN and total bilirubin ≤ 1.5 xULN (isolated predominantly indirect hyperbilirubinaemia due to Gilbert's syndrome is acceptable for inclusion)
5. ECOG Performance Status of 0, 1, or 2
6. Age ≥ 18 years
7. Life expectancy of at least 3 months
8. Signed written informed consent prior to performing any study-specific procedures

Main exclusion criteria:

1. Grade 3b follicular lymphoma or evidence that the indolent lymphoma has transformed to aggressive lymphoma as verified by biopsy confirmation [e.g. constitutional symptoms, poor performance status, fast growing tumour or increasing lactate dehydrogenase (LDH) level]
2. Previous allogeneic stem cell transplant
3. Previous external beam radiation therapy to the pelvis. Previous external beam radiation therapy for bony disease to the cranium, mediastinum, and axilla or to more than 3 vertebral bodies
4. More than 10 mg prednisolone daily at the time of randomisation
5. Prior bendamustine treatment within 1 year of randomisation not resulting in a CR or PR for at least 6 months
6. Known CNS involvement of indolent lymphoma
7. Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of definitively treated non-melanoma skin cancer, or successfully treated in situ carcinoma, are eligible
8. Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C
9. Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months of screening, congestive heart failure, and arrhythmia requiring therapy, with the exception of extrasystoles or minor conduction abnormalities. Subjects with well controlled congestive heart failure and atrial arrhythmias need not be excluded but should be discussed with the study Medical Monitor
10. Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease
11. History of significant cerebrovascular disease or event with significant symptoms or sequelae
12. Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator assessment)
13. Jaundice
14. Known HIV, Hepatitis B or Hepatitis C positive
15. Creatinine clearance ≤ 10 mL/min (measured or estimated using Cockcroft and Gault equation)
16. Treatment with any known non-marketed drug substance or experimental therapy within 5-terminal half-lives or 4 weeks prior to screening, whichever is longer or currently participating in any other interventional clinical study unless the sole purpose of the study is for collection of survival data
17. Known or suspected inability to comply with study protocol
18. Lactating women, women with a positive pregnancy test at screening or women (of childbearing potential) as well as men with partners of childbearing potential, who are not willing to use adequate contraception from study start through last treatment dose and for 6 months following cessation of treatment. Female contraception must be individually recommended by an expert. Adequate contraception is defined as abstinence, oral contraceptive, either combined or progestogen alone, injectable progestogen, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, intrauterine device (IUD) or intrauterine system (IUS), male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject, or double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository).

20.Major surgery less than 30 days prior to start of treatment. 21.Known hypersensitivity to the active substance or any excipients that cannot be controlled by appropriate pre-medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-02; Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 8 cycles of 21 days, then follow up every 3 months
  Screening of 14 days, prior to ramdomisation. 8 cycles of 21 days, then follow up every 3 months after end of last cycle until disease progression, then every 6 months.

SECONDARY OUTCOMES:
Overall Response Rate | 8 cycles of 21 days, then follow up every 3 months until progressive disease, then every 6 months for overall survival
  Complete remission (CR)/partial remission (PR), Duration of response (DR), Overall survival (OS), Safety and tolerability, Change in health related quality of life (HRQL) measures

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (2):
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide
- Dr Ludmila Demitrovicova, Bratislava, Slovakia